CLINICAL TRIAL: NCT02831621
Title: Effect of Diet Plus Exercise Versus Diet Alone on the Reduction of Ectopic Fat Deposition in Adults With Overweight
Brief Title: Exercise and Ectopic Fat Deposition
Acronym: ectofat
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universiteit Antwerpen (Other)
Responsible Party: Principal Investigator, Wendy Hens, candidate PHD, Universiteit Antwerpen
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 14/17/205
Record Dates: First submitted 2016-07-08; First posted 2016-07-13 (Estimated); Last update posted 2019-01-25 (Actual); Status verified 2019-01

CONDITIONS: Overweight
Keywords: overweight; ectopic fat; exercise; diet
MeSH Terms: conditions — Overweight; Motor Activity | interventions — Diet

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- diet (usual care) (Active Comparator): All participants will receive a hypocaloric diet based on the individual resting metabolic rate. Resting metabolic rate (RMR) will be estimated using the WHO formula or measured using indirect calorimetry. Total energy expenditure will be calculated by multiplying RMR with a physical activity level (PAL). The used physical activity level will be 1.3. A hypocaloric diet with an energy deficit of 500 kcal/day will be prescribed. Participants will see a skilled dietician two-weekly the first month and on a monthly basis the next five months to discuss problems and solutions or coping strategies. The first consultation will have a duration of 60 minutes, the next consultations will have a duration of approximately 30 minutes. Each visit, nutritional compliance will be recorded on a 0 to 10 numeric rating scale. The usual care group will be asked to continue with their normal physical activity during the six-month intervention period.
  Interventions: Behavioral: lifestyle intervention (diet OR diet+exercise)
- diet+exercise (Experimental): For participants of this group, usual care will be supplemented with a prescribed exercise program. For this exercise program the participants will be referred to a local fitness club near home, free of charge. Aerobic training will be done at an intensity of 90-95% of the heart rate achieved at the RCP. Aerobic training will have a duration of 30 to 45 minutes, according to the training stage. Cardio training will be performed on different cardio devices and strength training will be done on isotonic strength training devices. Each training day, core stability training will be completed with four strength exercises for large muscle groups. Each exercise will be done in two sets of 15 repetitions with the goal to achieve better muscular strength endurance.
  This combined training will be done individually during six months, three times/week.
  In this study, an effort is made to reach a uniform manner of guidance to the physical activity program.
  Interventions: Behavioral: lifestyle intervention (diet OR diet+exercise)

INTERVENTIONS:
Behavioral: lifestyle intervention (diet OR diet+exercise) — diet or diet+fitness training

SUMMARY:
Excess ectopic fat deposition is associated with development of cardiovascular and metabolic diseases. This study investigates how lifestyle interventions can have an effect on different sites of ectopic fat deposition and cardiovascular or metabolic factors. Moreover, the clinical and economic value of exercise to supplement a hypocaloric diet is investigated.

Endocrinologists of the University Hospital of Antwerp, Belgium, will be recruiting women during consultations. Also, recruitment posters will be used in the University Hospital of Antwerp and the University of Antwerp. Potential participants meeting all a priori set inclusion and exclusion criteria will be randomized by minimization method to a hypocaloric diet group (usual care) or a group of hypocaloric diet combined with physical fitness training. Both groups will undergo an intake procedure in which personal goals are set and barriers to changes in behavior will be discussed. Ectopic fat deposition will be measured by imaging techniques after three and six months of intervention. Based on the known relationship between ectopic fat and cardiovascular outcomes, the short term study results will then be extrapolated to an estimation of the reduction of cardiovascular events.

The following clinical outcomes will be presented: change in ectopic fat in the abdomen (visceral fat), the liver (intra hepatic lipids), skeletal muscle (intra myocellular lipids), heart (epicardial fat) after a dietary or combined (diet+physical activity) intervention. The impact of supervised exercise in addition to diet will be expressed in projected healthcare costs and quality adjusted life years.

DETAILED DESCRIPTION:
protocol of the study was published, Hens et al. (physioscience 2017; 13: 80-87)

ELIGIBILITY:
Inclusion Criteria:

* Participants should be willing to undergo a weight loss intervention and body weight must be stable during the past six months.
* There will be no upper eligibility criterion for body mass index (BMI) but BMI should be at least 27 kg/m².

Exclusion Criteria:

* Individuals who have a clinical history of type 2 diabetes, prediabetes (with use of medication), or hypothyroidism will be excluded.
* when postmenopausal; Premenopausal state will be verified by hormonal data (follicle-stimulation hormone (FSH) < 25 mU/ml and estradiol > 20 pg/ml).
* Subjects will not be allowed when pregnancy is planned
* when physical activity is not possible due to problems of the musculoskeletal system
* when changes in medication (e.g. beta blockers) are advised by an endocrinologist.
* when smoking
* when drinking more than two alcoholic consumptions/day or binge drinking (self-reported)
* when taking medication that influences body weight or metabolism (e.g. tricyclic antidepressants)
* Since all participants will undergo medical imaging, exclusion criteria related to MRI and CT scans are also applicable.

Ages: 18 Years to 60 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 60 (Actual)
Dates: Start 2016-06 (Actual); Primary Completion 2017-08 (Actual); Study Completion 2019-01 (Actual)

PRIMARY OUTCOMES:
hepatic lipid content | start - 3 months - 6 months - 12 months
  The hepatic lipid content will also be measured by a 3T MRI scanner (SIEMENS MAGNETOM Prisma, Siemens Healthcare AG, Zürich, Germany). The body coil will be positioned around the chest, as the subjects lay supine. MRI data will be acquired using STEAM, with the parameter setting as follows: 3.0 cm³ voxel in the right liver, TR/TE 3000/20 ms, and no water suppression.
intra myocellular lipids | start - 3 months - 6 months - 12 months
  1H-magnetic resonance spectroscopy (1H-MRs) will be used to quantify lipid levels in the tibialis anterior (slow-twitch) muscle of each subject.The right calf of each subject will be positioned near isocenter surrounded by a body coil within a 3T MRI scanner (SIEMENS MAGNETOM Prisma, Siemens Healthcare AG, Zürich, Germany) following manual shimming on the volume of interest to ensure maximum ﬁeld homogeneity. The 1H-MRs data will be acquired by a single-voxel Point-Resolved Spectroscopy (PRESS) acquisition. Imaging parameters will be set as follows; repetition time (TR)/echotime (TE) 2000/33 ms, voxel size 15 mm³, and weak water suppression.
pericardial and epicardial fat | start - 3 months - 6 months - 12 months
  Multislice ECG-triggered CT will be used to measure pericardial and epicardial fat areas. All scans will be performed at end-diastole and slice thickness of 2.5 mm. No contrast liquid will be used. Data will be analyzed using the corresponding workstation (GE, AW Volumeshare 2).
visceral fat | start - 3 months - 6 months - 12 months
  A single slice CT of the abdomen will be used to evaluate cross-sectional abdominal visceral adipose tissue areas at the L4-L5 region. The abdominal fat mass and its distribution in visceral adipose tissue (VAT) and subcutaneous adipose tissue (SAT) will be calculated by area measurement on the corresponding CT slice.
antropometric and metabolic parameters | start - (some at) 3 months - 6 months - 12 months
  Every participant will undergo a standard metabolic screening at the beginning of the study. This will include a detailed interview and a clinical examination with anthropometry.
health economic evaluation | start - 3 months - 6 months - 9 months - 12 months
  questionnaires will be used

CONTACTS AND LOCATIONS:
Locations (1):
- University Hospital of Antwerp, Antwerp, Belgium

REFERENCES:
- [Derived] Hens W, Vissers D, Annemans L, Gielen J, Van Gaal L, Taeymans J, Verhaeghe N. Health-related costs in a sample of premenopausal non-diabetic overweight or obese females in Antwerp region: a cost-of-illness analysis. Arch Public Health. 2018 Jul 30;76:42. doi: 10.1186/s13690-018-0285-1. eCollection 2018. PMID 30069308